CLINICAL TRIAL: NCT05224817
Title: Prospective, Multicenter Derivation and Validation of a NECROtizing Soft Tissue Infections (NECROSIS) Score
Brief Title: NECROtizing Soft Tissue Infections and Their Scoring System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 056.GME.2019.D
Record Dates: First submitted 2019-11-04; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Necrosis
MeSH Terms: conditions — Necrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Necrotizing soft tissue infections (NSTIs) — There will be no direct interaction with subjects and involves no interventions; study is conducted completely via review of electronic health records. Our site will only collect data from the Methodist Dallas Medical Center.

SUMMARY:
Primary Objective:

The primary objective of this study is to develop and validate a clinical risk index score for identifying NSTIs in emergency general surgery patients being evaluated for a severe skin and soft tissue infection.

Secondary Objectives:

To describe the contemporary microbiology of NSTIs and explore the effects on outcomes and to identify predictors of amputation and mortality.

DETAILED DESCRIPTION:
This study is designed as a multicenter, prospective, observational study. There will be no direct interaction with subjects and involves no interventions; study is conducted completely via review of electronic health records. Our site will only collect data from the Methodist Dallas Medical Center. We plan to complete the data collection and analysis by 12/30/2021.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age ≥18 years old and ≤89 years old) with suspected or confirmed NSTI

Exclusion Criteria:

* Age <18 years old and age > 89 years
* Pregnancy
* Prisoners
* Below ankle diabetic foot infections complicated by peripheral vascular disease
* Burn wounds

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: study is conducted completely via review of electronic health records. Our site will only collect data from the Methodist Dallas Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 1010 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in the presence of necrosis | up to 30 days
  presence of necrosis-"dishwater" fluid or deliquescent tissues
Change in the presence of necrosis | up to 30 days
  thrombosed vessels or absence of bleeding
mortality length of time in hospital | 30-90 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided